CLINICAL TRIAL: NCT04586998
Title: Prospective Multicenter Open-Label Single Group Study on the Comparison Between Propofol Concentration in Exhaled Breath and Blood Plasma Using the Propofol Monitor Edmon in Patients Undergoing Elective Surgery Under Total Intravenous Anaesthesia
Brief Title: Comparison Between Propofol Concentration in Exhaled Breath and Blood Plasma Using the Exhaled Drug Monitor "Edmon"
Acronym: ProDect
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HC-G-H-1716
Record Dates: First submitted 2020-09-18; First posted 2020-10-14 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Elective Surgical Procedures; Anesthesia, Intravenous
Keywords: EDMON; Propofol detection; Exhaled breath; Drug monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exhaled drug monitor "Edmon" (Experimental): Comparison between propofol in exhaled breath and blood plasma
  Interventions: Device: Exhaled drug monitor "Edmon"

INTERVENTIONS:
Device: Exhaled drug monitor "Edmon" — Taking samples of exhaled breath every minute during elective surgery in comparison to blood samples taken at predefined time points.

SUMMARY:
Edmon is the first Communauté Européenne (CE) marked medical device able to continuously measure propofol in the exhaled breath of patients under sedation or anaesthesia with propofol. Current scientific publications indicate that it makes sense from a pharmacologic point of view to measure propofol in the exhaled air.

If the present study can show the Edmon to be able to detect small differences in propofol plasma concentration it will underline the clinical value of measuring propofol in the exhaled breath. This might be an opportunity for a significant improvement in patient monitoring.

ELIGIBILITY:
* Inclusion criteria

  * Male or female patients undergoing elective surgical procedures
  * Expected duration of the surgical procedure > 1h
  * General anaesthesia (TIVA) with propofol and remifentanil under orotracheal intubation
  * Medical need for an arterial line for an invasive haemodynamic monitoring during anaesthesia
  * Written informed consent
  * Age ≥ 18 years
  * ASA I-III
  * BMI < 35 kg/m²
  * Women of child bearing potential: negative pregnancy test
  * BIS monitoring feasible (e.g. no surgical procedures on the frontal brain)
  * The patient is expected to be extubated in the OR after end of surgery
* Exclusion criteria

  * Patients with contraindications for propofol, remifentanil or for the planned anaesthetic procedure
  * Cardiac surgery
  * Lung surgery
  * Organ transplant procedures
  * Pulmonary diffusion anomalies (e.g. pulmonary fibrosis), known from medical history
  * Patients on renal replacement therapy
  * Participation in another interventional trial
  * Breastfeeding women
  * Unilateral lung ventilation
  * Emergency surgery
  * Patient is not able to give his/her written informed consent
  * Patients with a haemoglobin level below 10 g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Propofol measurements | During elective surgical procedure lasting longer than 1 hour
  To investigate the correlation between propofol concentrations in exhaled breath and blood plasma in patients undergoing elective surgical procedures under total intravenous anaesthesia.

SECONDARY OUTCOMES:
Identification of confounders with an impact on propofol exhaled breath concentration, e.g.among ventilatory and circulatory parameters | During elective surgical procedure lasting longer than 1 hour
  To identify confounders among ventilatory and circulatory parameters by correlating the course of propofol values with courses of single parameters from vital sign monitor or anaesthetic machine (e.g. systolic blood pressure or positive end-expiratory pressure (PEEP))
Evaluation of the correlation between propofol exhaled breath concentration and EEG index values | During elective surgical procedure lasting longer than 1 hour
  For that correlation EEG index values (Bispectral index (BIS) and suppression ratio) will be corrected by calculated remifentanil plasma concentration and then correlated to propofol exhaled breath concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Volk, Prof. Dr., Principal Investigator — Universitaetsklinikum des Saarlandes